CLINICAL TRIAL: NCT03694847
Title: Comparative Characteristics of Asthmatic Patients With and Without Nasal Polyposis: an Observational, Cross-sectional Study of the Quebec Heart and Lung Institute-Laval University Asthma Database.
Brief Title: Asthma With Nasal Polyposis
Status: Completed | Type: Observational
Sponsor: Louis-Philippe Boulet (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor-Investigator, Louis-Philippe Boulet, MD, FRCPC, FCCP, respirologist, Laval University
Organization: Laval University (Other)
Other Study IDs: CER21489
Record Dates: First submitted 2018-10-02; First posted 2018-10-03 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Asthma; Nasal Polyps
Keywords: asthma; chronic rhinosinusitis; nasal polyposis
MeSH Terms: conditions — Asthma; Nasal Polyps

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asthma with CRSwNP: Asthmatic patients with a diagnosis of CRSwNP
- Asthma without CRSwNP: Asthmatic patients without a diagnosis of CRSwNP

SUMMARY:
Asthma is often associated with various comorbidities that may influence its clinical expression. Among those, chronic rhinosinusitis with nasal polyposis (CRSwNP) is observed in 5% of cases. Asthmatic patients with CRSwNP appear to have more severe and poorly controlled asthma, as well as greater bronchial and systemic inflammation, especially those using inhaled corticosteroids as control medication. However, this remains to be validated. In the last decade, there has been interest labeled for phenotyping of asthma and CRSwNP. However, there is scarce data on the phenotype of asthma with CRSwNP.

This study aims to describe the phenotype of asthmatic patients with CRSwNP according to the clinical, physiological and inflammatory characteristics and whether there is a more severe phenotype related to the dose of inhaled corticosteroids and the percentage of induced sputum eosinophils.

DETAILED DESCRIPTION:
This study will compare the characteristics of asthmatic patients with CRSwNP with those without CRSwNP.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged 18 years and over 2. With a proven diagnosis of asthma as defined by one of the above criteria of current guidelines:

  1. Forced expiratory volume in one second (FEV1) increase by at least 12% (and ≥200 ml) after administration of a bronchodilator
  2. Current asthma symptoms and a methacholine provocative concentration inducing a 20% fall in FEV1 (PC20) <16 mg/ml
  3. A respirologist's current diagnosis of asthma found in the patient's medical report 3. Non-smokers or smokers/ex-smokers defined as someone with a smoking history <10 pack-years 4. Stable asthma and asthma medication for at least 4 weeks before data analysis 5. Written informed consent obtained for inclusion in the database

     Patients with CRSwNP

     1. With a proven diagnosis of CRSwNP, based on endoscopy and defined as the presence of endoscopically visible bilateral polyps growing from the middle meatus with or without involvement of the nasal cavities

     Exclusion Criteria:
     1. Any respiratory disease apart from asthma and CRSwNP
     2. Current or ex-smokers should not have a smoking history ≥10 pack-years before data analysis. Patients who administer nicotine in other forms (patches, chew tobacco, e-cigarette, etc.) will be excluded
     3. Unstable asthma medication <4 weeks before index date
     4. Asthma exacerbation (see definition below) <4 weeks before index date
     5. Respiratory tract infection <4 weeks before index date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asthmatic patients from the Quebec city region.
Sampling Method: Non-Probability Sample
Enrollment: 1293 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
Asthma severity | Baseline
  Prevalence of asthmatic with CRSwNP in mild, moderate and severe asthma

SECONDARY OUTCOMES:
Sputum inflammatory phenotype | Baseline
  Prevalence of patients with CRSwNP in each inflammatory sub groups: eosinophilic, neutrophilic, paucygranulocytic, Mix

CONTACTS AND LOCATIONS:
Overall Officials: Louis-Philippe Boulet, MD, Principal Investigator — IUCPQ-UL
Locations (1):
- Centre de recherche de l'Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Birs I, Boulay ME, Bertrand M, Cote A, Boulet LP. Heterogeneity of asthma with nasal polyposis phenotypes: A cluster analysis. Clin Exp Allergy. 2023 Jan;53(1):52-64. doi: 10.1111/cea.14247. Epub 2022 Nov 1. PMID 36317421